CLINICAL TRIAL: NCT02713724
Title: Effects of a Personalized Training Program on Trans-thoracic Adenosine-assisted Coronary Flow Reserve in Healthy Volunteers
Brief Title: Effects of Personalized Training Program on Coronary Flow Reserve in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Sara Svedlund, MD PhD, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GoteborgU_SSv
Record Dates: First submitted 2015-12-17; First posted 2016-03-21 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease; Heart Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Exercise; alpha,beta-diacryloxypropionic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAPS-group (Active Comparator): Physical exercise
  Interventions: Behavioral: physical exercise
- Standard-group (Active Comparator): Limited physical exercise
  Interventions: Behavioral: limited physical exercise

INTERVENTIONS:
Behavioral: physical exercise — DAPS-group will follow a personal adjusted training program including instructions from a personal trainer Standard-group will receive a membership at a gym but limited instructions
  Other Names: DAPS
  Arms: DAPS-group
Behavioral: limited physical exercise — The standard group will receive a membership at a gym but limited instructions and no access to a personal trainer
  Other Names: Standard
  Arms: Standard-group

SUMMARY:
This study investigates whether an individualized exercise program, including a personal trainer, can improve cardiovascular status quantified with ultrasound to assess coronary flow reserve and other non-invasive techniques. The subjects in the study will be divided into two groups; one group will have a personalized exercise- and nutrition program and the other group will have acess to a gym membership, but no personal trainer.

DETAILED DESCRIPTION:
Coronary heart disease is one of our most common diseases that causes significant morbidity and mortality. Because the risk of serious cardiovascular events, such as myocardial infarction and death, is evident in this patient population, it is of utmost importance to develop diagnostic methods to identify patients at risk. The most appropriate diagnostic methods are those that are safe to implement for both patient and physician, but also accessible and cost-efficient.

By using non-invasive techniques such as ultrasound, coronary artery function can be examined as coronary flow reserve (CFR). In the platform of non-invasive techniques used by the investigators for examinations of cardiovascular status, other methods are included, such as measurement of intima-media thickness in the carotid and radial arteries. The investigators goal is to compare the group with the personalized program with its placebo, and to compare the two study-groups with each other, to investigate whether the personalized program provides greater health benefits.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers
* no current medication,
* no known diseases that require regular medication
* no known risk factor for cardiovascular disease (hypertension, hyperlipidemia, diabetes, heredity, obesity, peripheral vascular disease)
* no physically fit athletes.

Exclusion Criteria:

* ongoing treatment with medicine containing dipyridamole (asasantin, persantin)
* known hypersensitivity to adenosine
* chronic obstructive pulmonary disease
* atrial fibrillation or other obvious arrythmias
* AV-block grade 2 or higher
* other serious illness

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve (CFR) | 3-6 months
  Ultrasound-assessed coronary flow reserve. Data will be presented as a ratio (no unit) between maximal mean hyperemia flow velocity and baseline velocity

SECONDARY OUTCOMES:
endothelial function | 3-6 months
  measured by EndoPath-device as RHI (reactive hyperemic index). Data will be presented as number of patients with abnormal RHI-values
cIMT (carotid artery intima-media thickness) | 3-6 months
  carotid artery intima-media thickness, data will be presented in mm
metabolic biomarkers | 3-6 months
  relevant metabolic blood biomarkers, data will be presented as numbers of participants with values of laboratory analyses below or above reference values
cardiovascular biomarkers | 3-6 months
  relevant cardiovascular blood biomarkers, data will be presented as numbers of participants with values of laboratory analyses below or above reference values
QoL (quality of life) | 3-6 months
  quality of life as measured by the validated scale PGWB (personal general well-being scale). Data will be presented as scores from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Svedlund, MD PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, VG-region, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westergren HU, Gan LM, Mansson M, Svedlund S. Randomized clinical trial studying effects of a personalized supervised lifestyle intervention program on cardiovascular status in physically inactive healthy volunteers. Oncotarget. 2018 Jan 3;9(10):9498-9511. doi: 10.18632/oncotarget.23958. eCollection 2018 Feb 6. PMID 29507706